CLINICAL TRIAL: NCT01615926
Title: Assessment of The Clinical Course of Dyspnea and Its Association With Respiratory Rate in Patients With Acute Heart Failure Syndromes
Brief Title: Assessment of The Clinical Course of Dyspnea in Acute Heart Failure Patients
Status: Terminated | Type: Observational
Why Stopped: Student related research project. Completion of allotted time.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Peter Pang, Associate Professor of Emergency Medicine, Northwestern University
Other Study IDs: MSSRP-IC2012
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Acute Heart Failure; Dyspnea
Keywords: dyspnea; shortness of breath; respiratory rate; orthopnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute heart failure (AHF) is defined as a gradual or rapid change in heart failure (HF) signs and symptoms, such as shortness of breath (also called dyspnea or breathlessness), leg swelling, fatigue, breathlessness with exertion, trouble sleeping flat at night, and weight gain resulting in a need for urgent therapy. AHF results in over 1 million hospitalizations every year, resulting in an enormous public health burden. Approximately 1/3rd of patients will either be re-hospitalized or die within three months, and the resultant financial costs are large. As such, improving outcomes for AHF patients is critically important. Shortness of breath is the most common reason why patients with AHF present to the ER. As such, understanding how severe this symptom is, how much it improves with current treatments is very important to both patients and physicians. The purpose of this study is to determine the degree to which your shortness of breath improves during the first few days of hospitalization and its association with how fast you are breathing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* AHFS is the primary working diagnosis for ER management and treatment with planned admission
* Have received IV diuretic therapy
* Enrolled within 3 hours of initial diuretic dose

Exclusion Criteria:

* BNP level is ≤ 300 pg/mL (may be initially enrolled and then will be excluded for second assessment)
* Transplant recipients of any kind
* Fever > 101.5
* Severe lung disease (required home O2 or daily oral steroids)
* Any ACS event within last 30 days
* Life expectancy less than 12 months for any reason
* Current treatment for any malignancy of any kind
* Cardiogenic shock and/or requiring IV inotropic therapy
* Pregnant or recently pregnant within last 90 days
* Inability to give appropriate written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who present to the Emergency Department with Acute Heart Failure
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine the association between respiratory rate and self-reported dyspnea in AHF patients. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Pang, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States